CLINICAL TRIAL: NCT03988959
Title: Surgical Management of Multiple Mucoepidermoid Carcinoma and Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Heba Sleem, professour doctor and principle investigator in department of oral and maxillofacial surgery, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110/2/2018
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Adenocarcinoma; Mucoepidermoid Carcinoma
Keywords: salivary gland tumor
MeSH Terms: conditions — Adenocarcinoma; Carcinoma, Mucoepidermoid; Salivary Gland Neoplasms

STUDY DESIGN:
Intervention Model Description: a case series was performed on 7 patients having mucoepidermoid carcinoma
Masking Description: No masking was done since its a case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control (Other): Standard resection
  Interventions: Procedure: resection of mucoeidermoid carcinoma

INTERVENTIONS:
Procedure: resection of mucoeidermoid carcinoma — Surgical resection parotid with preservation of facial nerve
  Other Names: Conservative superficial partoidectomy

SUMMARY:
A case series of patient having mucoepidermoid carcinoma, had standard treatment protocol and surgeries and followup was performed and the patient postoperative quality of life and recurrent rate was recorded

DETAILED DESCRIPTION:
This case series presents mucoepidermoid carcinoma. Palatal mass was resected with safety margin then immediate opturator inserted; superficial parotidectomy was also done for parotid lesion sparing facial nerve. Post-operative radiotherapy was recommended by pathologist due to evident perineural spread. The patient is tumor free after one year follow-up.

Clinical reports about synchronous multiple salivary tumors are very rare, consequently there is little known about its management and clinical presentation. Presence of one or more risk factor should favor expectation of multiple tumors and mandate examination of all salivary tissues. Each tumor should be diagnosed and treated separately according to its nature and extension.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from salivary gland tumor

Exclusion Criteria:

* healthy patients with no tumors

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Quality of life | 6 months
  in grades the quality of life of patients is assessed by visual analogue scale in a scale from 1-10. higher values indicates better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Diaa, Prof Dr, Study Director — Dean of Faculty
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
No plan to share those data currently with other researchers